CLINICAL TRIAL: NCT02255136
Title: An Evidence-based Single-blind Randomized Controlled Trial Searching for the Efficacy of Homoeopathic Medicines in Reducing Serum Levels of Cytokines (IL - 10, 13) and Immunoglobulin E in Allergic Rhinitis and/or Induced Bronchial Asthma
Brief Title: Efficacy Study of Homeopathic Medicines in Treatment of Allergic Rhinitis and/or Induced Bronchial Asthma
Acronym: SBRCTHILARBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahesh Bhattacharyya Homoeopathic Medical College and Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Shubhamoy Ghosh, MD (Hom), Lecturer of the Department of Pathology & Microbiology, Mahesh Bhattacharyya Homoeopathic Medical College and Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 793/MBHMCH/CH/Adm/01/2011; CTRI/2012/02/002419 (Registry Identifier: Clinical Trial Registry - India)
Record Dates: First submitted 2012-02-15; First posted 2014-10-02 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Rhinitis; Allergic, With Asthma
Keywords: Interleukin; Immunoglobulin; Homeopathy; Allergic Rhinitis; Asthma
MeSH Terms: conditions — Rhinitis; Rhinitis, Allergic; Asthma

STUDY DESIGN:
Intervention Model Description: Prospective, single-blind (subject), randomized, placebo-controlled, parallel group, interventional clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individualized homeopathic medicines (Experimental): Psorinum, Tuberculinum, Medorrhinum, Calcarea carbonica, Natrum sulphuricum etc. as indicated; Rescue medicines, e.g. Aralea racemosa, Arsenicum album, Histamine hydrochloride, House dust, Ipecacuanha, Antimonium tartaricum, Grindelia robusta etc. as indicated; 5 ml dose of indicated homeopathic medicine in centesimal or 50 millesimal potencies as appropriate; administered twice daily for 1 year
  Interventions: Other: Individualized homeopathic medicines
- Intervention placebo (Placebo Comparator): 5 ml dose made up of single drop of rectified spirit in 5 ml distilled water, identical in appearance of homeopathic medicine, to be administered twice daily for 1 year
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Individualized homeopathic medicines — 5 ml dose of indicated individualized homeopathic medicine in centesimal or 50 millesimal potencies as appropriate; twice daily for 1 year
  Arms: Individualized homeopathic medicines
Other: Placebo — Placebo, in the form of a single drop of rectified spirit in 5 ml of distilled water
  Other Names: Placebo: distilled water
  Arms: Intervention placebo

SUMMARY:
The purpose of this study is to test whether individualized homeopathic medicines can produce any significant effect beyond placebo in treatment of allergic rhinitis and/or induced bronchial asthma

DETAILED DESCRIPTION:
A prospective, single-blind (subject), randomized, placebo-controlled, parallel group, interventional clinical trial is being conducted on 100 participants (subjects 50, control 50) suffering from allergic rhinitis and/or induced bronchial asthma since March 1, 2012 at Mahesh Bhattacharyya Homeopathic Medical College and Hospital, Government of West Bengal. This trial is aimed at exploring the efficacy of homeopathic medicines in comparison with placebo in reducing serum interleukin 10, 13 and immunoglobulin E measured at timeline of 1 year of treatment and absolute eosinophil count every 4 months up to 1 year. Matching for independent and consequent variables will be done to test for bias. Parametric or non-parametric tests will be employed as per distribution of data at the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 and 65 years
* Both sexes
* Atopic: reactive to allergens with positive skin prick test (SPT) results and/or eosinophilia
* More than 1 year history of allergic rhinitis and/or induced bronchial asthma

Exclusion Criteria:

* Nasal abnormalities causing obstruction, e.g. nasal polyp(s), deviated septum etc.
* Previous homoeopathic immunotherapy for allergic rhinitis
* Allergen avoidance in past 6 weeks
* Away from usual environment for more than 1 week during trial
* Severe asthma cases as detected clinically
* Respiratory infection
* Severe concomitant disease
* Pregnancy, breast feeding, or likelihood of pregnancy
* Oral or parenteral steroids and/or decongestant in past 6 months
* Conventional desensitization in past 3 months

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Serum Interleukin 10 and 13 level | 1 year

SECONDARY OUTCOMES:
Incidence of adverse events if any | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shubhamoy Ghosh, MD(Hom), Principal Investigator — Lecturer of the Department of Pathology & Microbiology
Locations (1):
- Mahesh Bhattacharyya Homeopathic Medical College & Hospital, Howrah, West Bengal, India

IPD SHARING:
Plan to Share IPD: Undecided